CLINICAL TRIAL: NCT00875147
Title: Impact of Pre-operative Bevacizumab on Complications After Resection of Colorectal Liver Metastases A Case Matched Control Study
Brief Title: Impact of Pre-operative Bevacizumab on Complications After Resection of Colorectal Liver Metastases
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ksenija Slankamenac, MD, University of Zurich
Other Study IDs: StV 12-2009
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Liver Metastases
Keywords: neoadjuvant chemotherapy; bevacizumab
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- with bevacizumab: Neoadjuvant chemotherapy with bevacizumab
  Interventions: Drug: bevacizumab
- without Bevacizumab: Neoadjuvant chemotherapy without Bevacizumab

INTERVENTIONS:
Drug: bevacizumab — Neoadjuvant chemotherapy with bevacizumab
  Groups: with bevacizumab

SUMMARY:
Hypothesis of the study: Neoadjuvant chemotherapy with Bevacizumab impairs postoperative outcome after resection of colorectal liver metastases.

DETAILED DESCRIPTION:
Bevacizumab is a humanized monoclonal antibody against vascular endothelial growth factor (VEGF) increasingly added to other drugs in the treatment of colorectal cancer. Bev is typically used in combination with other chemotherapeutic agents such as oxaliplatin, irinotecan, leucovorin and 5-fluorouracil (5-FU) for treatment of patients with CRLM. The objective of this study was to assess the impact of neoadjuvant bevacizumab on clinical outcome after hepatectomy of colorectal liver metastases (CRLM).

Patients, who underwent liver resection due to colorectal liver metastases after neoadjuvant chemotherapy, operated between 2005 and 2007 will be evaluated retrospectively. The patients will be distributed in two groups, either with or without bevacicumab. Outcome parameters are mortality, complications, hospital stay and ICU stay. To increase the power of the study the total number of patients will be increased by adding patients from other centers. Results will be adjusted for the propensity of developing complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neoadjuvant chemotherapy prior to liver resection

Exclusion Criteria:

* Patients without neoadjuvant chemotherapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who underwent liver resection due to CRLM between 2005 and 2007, were retrospectively assessed for eligibility. Patients with chemotherapy containing Bev prior to surgery are identified consequtively. This group of patient with preoperative Bev is matched to patients without Bev. Consecutive patients with neoadjuvant application of Bevacizumab will be matched to patients without Bevacizumab. Results are statistically adjusted according to potential confounders.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Overall complications | postoperative

SECONDARY OUTCOMES:
specific complications such as liver insufficiency, length of hospital stay | postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Breitenstein, MD, Principal Investigator — Departement of Visceral and Transplantation Surgery of University hospital of Zurich
Locations (3):
- Centre de Chirurgie Viscérale et de Transplantation, Hautepierre Hospital, Strasbourg, Strasbourg, France
- Division of hepato-biliary-pancreatic surgery. Department of surgery, "Josep Tureta" Hospital, Girona, Girona, Spain
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland